CLINICAL TRIAL: NCT05977881
Title: Impact of a Novel HIV Peer Navigation and Overdose Prevention Intervention on Engagement in the HIV Prevention and Treatment Cascade
Brief Title: Substance Checking Outreach and Pre-Exposure Prophylaxis (PrEP) Engagement Study
Acronym: SCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Baltimore City Health Department (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00017498; 5R01DA053184 (NIH)
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections
Keywords: Drug Use; Overdose; PrEP; Harm Reduction
MeSH Terms: conditions — HIV Infections; Drug Overdose; Harm Reduction

STUDY DESIGN:
Intervention Model Description: The study interventional model is at the community level; the intervention will be offered in all areas in which the cohort will be recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SCOPE Cohort (Other): A cohort of PWUD (N=500) living in Baltimore. We will follow-up with participants every 6 months (for 18 months) in five recruitment zones throughout Baltimore (n=125/zone). The four recruitment zones will overlap the intervention sites. There will be four study visits (baseline, 6 months, 12 months, 18 months) total for participants.
  Interventions: Other: CHECKIT!

INTERVENTIONS:
Other: CHECKIT! — Participants will not be assigned to the intervention as it will be available to everyone.
  Check it will be a van-based HIV- and overdose-prevention program offered in the four areas of Baltimore city from which study participants are recruited. Intervention services will include point-of-care drug checking and PrEP assessment, prescription, and management, and they will be available to everyone, regardless of whether they are part of the SCOPE study cohort or not.
  Individual-level service usage data collected by intervention staff will not be considered in analysis of outcomes. However, study participants will self-report Check it utilization on the internally-developed surveys at 6, 12, and 18 months.

SUMMARY:
Through the proposed Substance Checking Outreach and Pre-Exposure Prophylaxis (PrEP) Engagement (SCOPE) study, the investigators will design and evaluate an overdose prevention and HIV prevention study among people who use drugs (PWUD). Specifically, SCOPE will provide access to drug-checking services for PWUD to better understand the contents of the drug supply, in combination with PrEP for those who are HIV-, to both reduce overdose and HIV among PWUD in Baltimore City.

DETAILED DESCRIPTION:
specific study aims are:

1. To prepare the drug-checking technology for deployment in the community through a three-phase process.

   1. To calibrate drug-checking technology through testing samples of illicit substances on the Bruker Alpha obtained from the Baltimore Police crime lab (N=335) and those obtained through the SPARC outreach sessions (N=100).
   2. To validate the drug-checking technology, measuring sensitivity and specificity in detecting illicit substances of public health relevance, by testing samples obtained through partnerships through Baltimore-based harm reduction organizations and comparing findings to the gold standard (laboratory testing).
   3. To pilot the study Bruker Alpha Fourier Transform Infrared Spectroscopy (FT-IR) drug checking machine among People who use drugs (PWUD) (N=20).
2. To develop a community-level, mobile, integrated drug checking and PrEP intervention aimed to increase PWUD engagement in the PrEP care continuum and reduce the burden of overdose.
3. To recruit a longitudinal cohort of people who use drugs (N=500) and follow-up at 6-month intervals for 18 months.
4. To implement the intervention and evaluate its impact on engagement in PrEP care (primary outcome) and overdose prevention among PWUD.

   1. To determine the incremental cost-effectiveness of the intervention in terms of HIV cases averted among PWUD.

The initial nonhuman subjects research plan focused on Aim's 1 drug checking machine calibration among samples procured from the Baltimore Police Forensics Lab tested in Dr. William Clarke's lab and from individuals interacting with SPARC staff during the outreach which occurs 3-4 times per week. These activities are referred to as "Phase 1" throughout this research plan. Based on emerging best practices and in consultation with other drug checking initiatives nationwide, the investigators have now expanded Aim 1 of the study to include three steps needed to prepare the machine for deployment in the field: The first (1a) was calibration of the machine to the local drug supply, as described above; the second (1b) which the investigators are adding in this amendment is an additional validation of the machine's functionality and comparison with gold standard technology; and the third (1c) is piloting the machine with 20 PWUD prior to rolling it out citywide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older,
* self-reports having used illicit stimulants or opioids at least once in the past 3 months,
* self-reports being HIV negative
* reports injection drug use in the past 6 months OR reports at least one of the following indicators of sexual HIV risk exposure in the past 6 months:

  1. Sexually Transmitted Infection (STI) diagnosis in the past 6 months
  2. "Condom-less" vaginal or anal sex in the past 6 months
* Willing to provide a urine sample for urine drug screening of substances
* Willing to undergo rapid HIV testing
* Willing to undergo STI testing

Exclusion Criteria:

* Determined to be too high or drunk or cognitively impaired, less than 18 years of age
* unwilling to provide all required biological specimens (Phase 3 only)
* unwilling/unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Current PrEP status as assessed by study team instrument items | Measured at Baseline, 6, 12, and 18 months
  Investigators will measure current PrEP status by assessing participant self-report using an internally developed questionnaire. Change in current PrEP status will be measured using three survey items asking participants 1) if they are currently prescribed either form of PrEP (pill form or injection), 2) currently taking/not taking the prescription, and 3) which type/brand of PrEP are they currently taking. The response range options for current prescription and currently taking PrEP are binary (yes/no) and nominal (choices) for type of PrEP prescribed. Participants will indicate whether they are currently prescribed PrEP, currently taking PrEP and which type prescribed/taking at each study visit.
Change in PrEP uptake as assessed by study team instrument items | Measured at 6, 12, 18 months
  Change in PrEP status (uptake) at follow-up is measured using three items with response range options for current prescription and currently taking PrEP are binary (yes/no) and nominal (choices) for type of PrEP prescribed. If participants self-report current PrEP use at follow-up, investigators will confirm the biological presence of PrEP using dried blood spot (DBS) sampling. Samples will be transported to the Clinical Pharmacology Analytical Laboratory (CPAL) where they will be processed using FDA-validated assays analyzing drug and metabolite concentrations. Sample results will be used to compare participant self-report on the study team survey instrument (e.g., what is the concordance/discordance between PrEP presence in DBS samples and yes/no responses to the currently taking PrEP survey item).

SECONDARY OUTCOMES:
Change in HIV Risk Behaviors as assessed by study team instrument items | Measured at Baseline, 6, 12, 18 months
  Investigators will measure change in HIV risk behaviors using self-report with an internally developed questionnaire; there are several items in the instrument to capture 1) episodes of syringe sharing in the prior 30 days and 2) episodes of unprotected vaginal or anal intercourse. Response options for HIV risk behaviors are continuous (counts # of times of episodes) and response options for HIV prevention techniques used are nominal; e.g., 'used a condom with my main sexual partner', or 'take HIV PrEP', or, 'did you use syringes after someone else?'.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Sherman, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Project de-identified IPD will made available for published analyses upon request. The investigators will also include the study protocol (IPD supporting information).
Supporting Information: Study Protocol
Time Frame: The time frame is for the project's IPD/supporting information is 'Unending'; the investigators will consider requests for data related to the project up to five years after publication.
Access Criteria: To access project IPD and supporting information, the investigators will consider requests for data from other researchers (university or governmental). The PI will review all requests, approve, and provide IPD access when appropriate.

REFERENCES:
- [Background] Murphy SL, Xu J, Kochanek KD, Arias E. Mortality in the United States, 2017. NCHS Data Brief. 2018 Nov;(328):1-8. PMID 30500322
- [Background] Hedegaard H, Minino AM, Warner M. Drug Overdose Deaths in the United States, 1999-2017. NCHS Data Brief. 2018 Nov;(329):1-8. PMID 30500323
- [Background] Centers for Disease Control and Prevention. HIV Infection Risk, Prevention, and Testing Behaviors among Persons Who Inject Drugs-National HIV Behavioral Surveillance: Injection Drug Use, 23 U.S. Cities, 2018. HIV Surveillance Special Report. 2020;24.
- [Background] Des Jarlais DC, Nugent A, Solberg A, Feelemyer J, Mermin J, Holtzman D. Syringe Service Programs for Persons Who Inject Drugs in Urban, Suburban, and Rural Areas - United States, 2013. MMWR Morb Mortal Wkly Rep. 2015 Dec 11;64(48):1337-41. doi: 10.15585/mmwr.mm6448a3. PMID 26655918
- [Background] Beyrer C, Malinowska-Sempruch K, Kamarulzaman A, Kazatchkine M, Sidibe M, Strathdee SA. Time to act: a call for comprehensive responses to HIV in people who use drugs. Lancet. 2010 Aug 14;376(9740):551-63. doi: 10.1016/S0140-6736(10)60928-2. PMID 20650515
- [Background] Aspinall EJ, Nambiar D, Goldberg DJ, Hickman M, Weir A, Van Velzen E, Palmateer N, Doyle JS, Hellard ME, Hutchinson SJ. Are needle and syringe programmes associated with a reduction in HIV transmission among people who inject drugs: a systematic review and meta-analysis. Int J Epidemiol. 2014 Feb;43(1):235-48. doi: 10.1093/ije/dyt243. Epub 2013 Dec 27. PMID 24374889
- [Background] Glick SN, Prohaska SM, LaKosky PA, Juarez AM, Corcorran MA, Des Jarlais DC. The Impact of COVID-19 on Syringe Services Programs in the United States. AIDS Behav. 2020 Sep;24(9):2466-2468. doi: 10.1007/s10461-020-02886-2. No abstract available. PMID 32333209
- [Background] Alpren C, Dawson EL, John B, Cranston K, Panneer N, Fukuda HD, Roosevelt K, Klevens RM, Bryant J, Peters PJ, Lyss SB, Switzer WM, Burrage A, Murray A, Agnew-Brune C, Stiles T, McClung P, Campbell EM, Breen C, Randall LM, Dasgupta S, Onofrey S, Bixler D, Hampton K, Jaeger JL, Hsu KK, Adih W, Callis B, Goldman LR, Danner SP, Jia H, Tumpney M, Board A, Brown C, DeMaria A Jr, Buchacz K. Opioid Use Fueling HIV Transmission in an Urban Setting: An Outbreak of HIV Infection Among People Who Inject Drugs-Massachusetts, 2015-2018. Am J Public Health. 2020 Jan;110(1):37-44. doi: 10.2105/AJPH.2019.305366. Epub 2019 Nov 14. PMID 31725317
- [Background] Atkins A, McClung RP, Kilkenny M, Bernstein K, Willenburg K, Edwards A, Lyss S, Thomasson E, Panneer N, Kirk N, Watson M, Adkins E, DiNenno E, Hogan V, Neblett Fanfair R, Napier K, Ridpath AD, Perdue M, Chen M, Surtees T, Handanagic S, Wood H, Kennebrew D, Cohn C, Sami S, Eubank S, Furukawa NW, Rose B, Thompson A, Spadafora L, Wright C, Balleydier S, Broussard D, Reynolds P, Carnes N, Haynes N, Sapiano T, McBee S, Campbell E, Batdorf S, Scott M, Boltz M, Wills D, Oster AM. Notes from the Field: Outbreak of Human Immunodeficiency Virus Infection Among Persons Who Inject Drugs - Cabell County, West Virginia, 2018-2019. MMWR Morb Mortal Wkly Rep. 2020 Apr 24;69(16):499-500. doi: 10.15585/mmwr.mm6916a2. No abstract available. PMID 32324723
- [Background] Strathdee SA, Beyrer C. HIV Outbreak in Indiana. N Engl J Med. 2015 Oct;373(14):1380-1. doi: 10.1056/NEJMc1510396. No abstract available. PMID 26422741
- [Background] Geddes L, Iversen J, Memedovic S, Maher L. Intravenous fentanyl use among people who inject drugs in Australia. Drug Alcohol Rev. 2018 Apr;37 Suppl 1:S314-S322. doi: 10.1111/dar.12668. Epub 2018 Feb 6. PMID 29405465
- [Background] Lambdin BH, Bluthenthal RN, Zibbell JE, Wenger L, Simpson K, Kral AH. Associations between perceived illicit fentanyl use and infectious disease risks among people who inject drugs. Int J Drug Policy. 2019 Dec;74:299-304. doi: 10.1016/j.drugpo.2019.10.004. Epub 2019 Nov 13. PMID 31733979
- [Background] Centers for Disease Control and Prevention. Preexposure prophylaxis for the prevention of HIV infection in the United States-2014: a clinical practice guideline. Atlanta: Centers for Disease Control and Prevention. 2014:67.
- [Background] Shrestha R, Copenhaver M. Exploring the Use of Pre-exposure Prophylaxis (PrEP) for HIV Prevention Among High-Risk People Who Use Drugs in Treatment. Front Public Health. 2018 Jul 13;6:195. doi: 10.3389/fpubh.2018.00195. eCollection 2018. PMID 30062091
- [Background] Centers for Disease Control and Prevention. HIV Infection Risk, Prevention, and Testing Behaviors among Persons Who Inject Drugs-National HIV Behavioral Surveillance: Injection Drug Use, 23 U.S. Cities, 2018. 2020;24:43.
- [Background] Bazzi AR, Biancarelli DL, Childs E, Drainoni ML, Edeza A, Salhaney P, Mimiaga MJ, Biello KB. Limited Knowledge and Mixed Interest in Pre-Exposure Prophylaxis for HIV Prevention Among People Who Inject Drugs. AIDS Patient Care STDS. 2018 Dec;32(12):529-537. doi: 10.1089/apc.2018.0126. Epub 2018 Oct 11. PMID 30311777
- [Background] Allen ST, O'Rourke A, White RH, Smith KC, Weir B, Lucas GM, Sherman SG, Grieb SM. Barriers and Facilitators to PrEP Use Among People Who Inject Drugs in Rural Appalachia: A Qualitative Study. AIDS Behav. 2020 Jun;24(6):1942-1950. doi: 10.1007/s10461-019-02767-3. PMID 31853771
- [Background] Jo Y, Bartholomew TS, Doblecki-Lewis S, Rodriguez A, Forrest DW, Tomita-Barber J, Oves J, Tookes HE. Interest in linkage to PrEP among people who inject drugs accessing syringe services; Miami, Florida. PLoS One. 2020 Apr 16;15(4):e0231424. doi: 10.1371/journal.pone.0231424. eCollection 2020. PMID 32298320
- [Background] Kuo I, Olsen H, Patrick R, Phillips G 2nd, Magnus M, Opoku J, Rawls A, Peterson J, Hamilton F, Kharfen M, Greenberg A. Willingness to use HIV pre-exposure prophylaxis among community-recruited, older people who inject drugs in Washington, DC. Drug Alcohol Depend. 2016 Jul 1;164:8-13. doi: 10.1016/j.drugalcdep.2016.02.044. Epub 2016 Mar 15. PMID 27177804
- [Background] Sherman SG, Schneider KE, Park JN, Allen ST, Hunt D, Chaulk CP, Weir BW. PrEP awareness, eligibility, and interest among people who inject drugs in Baltimore, Maryland. Drug Alcohol Depend. 2019 Feb 1;195:148-155. doi: 10.1016/j.drugalcdep.2018.08.014. Epub 2018 Oct 22. PMID 30639794
- [Background] Walters SM, Rivera AV, Starbuck L, Reilly KH, Boldon N, Anderson BJ, Braunstein S. Differences in Awareness of Pre-exposure Prophylaxis and Post-exposure Prophylaxis Among Groups At-Risk for HIV in New York State: New York City and Long Island, NY, 2011-2013. J Acquir Immune Defic Syndr. 2017 Jul 1;75 Suppl 3:S383-S391. doi: 10.1097/QAI.0000000000001415. PMID 28604443
- [Background] Stein M, Thurmond P, Bailey G. Willingness to use HIV pre-exposure prophylaxis among opiate users. AIDS Behav. 2014 Sep;18(9):1694-700. doi: 10.1007/s10461-014-0778-z. PMID 24752703
- [Background] McFarland W, Lin J, Santos GM, Arayasirikul S, Raymond HF, Wilson E. Low PrEP Awareness and Use Among People Who Inject Drugs, San Francisco, 2018. AIDS Behav. 2020 May;24(5):1290-1293. doi: 10.1007/s10461-019-02682-7. PMID 31563984
- [Background] Roth A, Tran N, Piecara B, Welles S, Shinefeld J, Brady K. Factors Associated with Awareness of Pre-exposure Prophylaxis for HIV Among Persons Who Inject Drugs in Philadelphia: National HIV Behavioral Surveillance, 2015. AIDS Behav. 2019 Jul;23(7):1833-1840. doi: 10.1007/s10461-018-2293-0. PMID 30267367
- [Background] Escudero DJ, Kerr T, Wood E, Nguyen P, Lurie MN, Sued O, Marshall BD. Acceptability of HIV Pre-exposure Prophylaxis (PREP) Among People Who Inject Drugs (PWID) in a Canadian Setting. AIDS Behav. 2015 May;19(5):752-7. doi: 10.1007/s10461-014-0867-z. PMID 25086669
- [Background] Mayer KH, Agwu A, Malebranche D. Barriers to the Wider Use of Pre-exposure Prophylaxis in the United States: A Narrative Review. Adv Ther. 2020 May;37(5):1778-1811. doi: 10.1007/s12325-020-01295-0. Epub 2020 Mar 30. PMID 32232664
- [Background] Walters SM, Reilly KH, Neaigus A, Braunstein S. Awareness of pre-exposure prophylaxis (PrEP) among women who inject drugs in NYC: the importance of networks and syringe exchange programs for HIV prevention. Harm Reduct J. 2017 Jun 29;14(1):40. doi: 10.1186/s12954-017-0166-x. PMID 28662716
- [Background] Roth AM, Aumaier BL, Felsher MA, Welles SL, Martinez-Donate AP, Chavis M, Van Der Pol B. An Exploration of Factors Impacting Preexposure Prophylaxis Eligibility and Access Among Syringe Exchange Users. Sex Transm Dis. 2018 Apr;45(4):217-221. doi: 10.1097/OLQ.0000000000000728. PMID 29465703
- [Background] Hershow RB, Gonzalez M, Costenbader E, Zule W, Golin C, Brinkley-Rubinstein L. Medical Providers and Harm Reduction Views on Pre-Exposure Prophylaxis for HIV Prevention Among People Who Inject Drugs. AIDS Educ Prev. 2019 Aug;31(4):363-379. doi: 10.1521/aeap.2019.31.4.363. PMID 31361517
- [Background] Beletsky L, Davis CS. Today's fentanyl crisis: Prohibition's Iron Law, revisited. Int J Drug Policy. 2017 Aug;46:156-159. doi: 10.1016/j.drugpo.2017.05.050. Epub 2017 Jul 18. PMID 28735773
- [Background] Mattson CL, Tanz LJ, Quinn K, Kariisa M, Patel P, Davis NL. Trends and Geographic Patterns in Drug and Synthetic Opioid Overdose Deaths - United States, 2013-2019. MMWR Morb Mortal Wkly Rep. 2021 Feb 12;70(6):202-207. doi: 10.15585/mmwr.mm7006a4. PMID 33571180
- [Background] Wilson N, Kariisa M, Seth P, Smith H 4th, Davis NL. Drug and Opioid-Involved Overdose Deaths - United States, 2017-2018. MMWR Morb Mortal Wkly Rep. 2020 Mar 20;69(11):290-297. doi: 10.15585/mmwr.mm6911a4. PMID 32191688
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857
- [Background] O'Donnell J, Gladden RM, Mattson CL, Kariisa M. Notes from the Field: Overdose Deaths with Carfentanil and Other Fentanyl Analogs Detected - 10 States, July 2016-June 2017. MMWR Morb Mortal Wkly Rep. 2018 Jul 13;67(27):767-768. doi: 10.15585/mmwr.mm6727a4. No abstract available. PMID 30001560
- [Background] Maryland Department of Health. Unintentional drug- and alcohol-related intoxication deaths in Maryland annual report 2017. Annapolis, Maryland. 2017.
- [Background] Drug Enforcement Agency. National Heroin Threat Assessment Summary - Updated. United States Drug Enforcement Administration;2016. DEA-DCT-DIR-031-16.
- [Background] Brunt TM, Nagy C, Bucheli A, Martins D, Ugarte M, Beduwe C, Ventura Vilamala M. Drug testing in Europe: monitoring results of the Trans European Drug Information (TEDI) project. Drug Test Anal. 2017 Feb;9(2):188-198. doi: 10.1002/dta.1954. Epub 2016 Feb 17. PMID 26888408
- [Background] Harper L, Powell J, Pijl EM. An overview of forensic drug testing methods and their suitability for harm reduction point-of-care services. Harm Reduct J. 2017 Jul 31;14(1):52. doi: 10.1186/s12954-017-0179-5. PMID 28760153
- [Background] Peiper NC, Clarke SD, Vincent LB, Ciccarone D, Kral AH, Zibbell JE. Fentanyl test strips as an opioid overdose prevention strategy: Findings from a syringe services program in the Southeastern United States. Int J Drug Policy. 2019 Jan;63:122-128. doi: 10.1016/j.drugpo.2018.08.007. Epub 2018 Oct 3. PMID 30292493
- [Background] Bardwell G, Kerr T. Drug checking: a potential solution to the opioid overdose epidemic? Subst Abuse Treat Prev Policy. 2018 May 25;13(1):20. doi: 10.1186/s13011-018-0156-3. PMID 29801458
- [Background] Sherman SG, Park JN, Glick J, et al. FORECAST Study Summary Report. Johns Hopkins Bloomberg School of Public Health. 2018.
- [Background] Sherman SG, Morales KB, Park JN, McKenzie M, Marshall BDL, Green TC. Acceptability of implementing community-based drug checking services for people who use drugs in three United States cities: Baltimore, Boston and Providence. Int J Drug Policy. 2019 Jun;68:46-53. doi: 10.1016/j.drugpo.2019.03.003. Epub 2019 Apr 13. PMID 30991301
- [Background] Morales KB, Park JN, Glick JL, Rouhani S, Green TC, Sherman SG. Preference for drugs containing fentanyl from a cross-sectional survey of people who use illicit opioids in three United States cities. Drug Alcohol Depend. 2019 Nov 1;204:107547. doi: 10.1016/j.drugalcdep.2019.107547. Epub 2019 Aug 23. PMID 31536877
- [Background] Rouhani S, Park JN, Morales KB, Green TC, Sherman SG. Harm reduction measures employed by people using opioids with suspected fentanyl exposure in Boston, Baltimore, and Providence. Harm Reduct J. 2019 Jun 24;16(1):39. doi: 10.1186/s12954-019-0311-9. PMID 31234942
- [Background] Gale NK, Heath G, Cameron E, Rashid S, Redwood S. Using the framework method for the analysis of qualitative data in multi-disciplinary health research. BMC Med Res Methodol. 2013 Sep 18;13:117. doi: 10.1186/1471-2288-13-117. PMID 24047204
- [Background] Biello KB, Bazzi AR, Vahey S, Harris M, Shaw L, Brody J. Delivering Preexposure Prophylaxis to People Who Use Drugs and Experience Homelessness, Boston, MA, 2018-2020. Am J Public Health. 2021 Jun;111(6):1045-1048. doi: 10.2105/AJPH.2021.306208. PMID 33950728
- [Background] Mistler CB, Copenhaver MM, Shrestha R. The Pre-exposure Prophylaxis (PrEP) Care Cascade in People Who Inject Drugs: A Systematic Review. AIDS Behav. 2021 May;25(5):1490-1506. doi: 10.1007/s10461-020-02988-x. PMID 32749627
- [Derived] Schneider KE, Nestadt DF, Martin EM, Morris M, Rouhani S, Weir BW, Sherman SG. Substance Checking Outreach and PrEP Engagement (SCOPE) Study: protocol for a non-randomised clinical trial in Baltimore, Maryland USA. BMJ Open. 2025 Jul 17;15(7):e101380. doi: 10.1136/bmjopen-2025-101380. PMID 40675636
- See also: National Institutes of Health. Substance Use Disorders Linked to Covid-19 Susceptibility — https://www.nih.gov/news-events/news-releases/substance-use-disorders-linked-covid-19-susceptibility